CLINICAL TRIAL: NCT06109727
Title: Acute Effect of tDCS on Motor Performance, Autonomic Control and Attentional and Executive Functions in Young Individuals
Brief Title: Acute Effect of tDCS in Young Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Taís Malysz, Professora, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 71695023.3.0000.5347
Record Dates: First submitted 2023-10-16; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the intervention group, the anodic stimulations will start after a ramp period of 30 s, followed by 20 min at 2 mili ampere and will end with a ramp of 30 s.
  Interventions: Device: cerebellar transcranial electrical stimulation
- Placebo (Placebo Comparator): In the simulated configuration, the ramp of 30 s will be immediately followed by the ramp of 30 s and without any current (Sham Group)
  Interventions: Device: cerebellar transcranial electrical stimulation

INTERVENTIONS:
Device: cerebellar transcranial electrical stimulation — Cerebellar transcranial electrical stimulation - 20 mA - 20 min

SUMMARY:
The aim of this study is to investigate the effect of transcranial electrical stimulation (tDCS) on motor performance, autonomic control and attentional and executive functions in young individuals.

DETAILED DESCRIPTION:
Gait research in young and healthy individuals increases knowledge about the neuromuscular structures involved in this motor act and thus helps to develop or adapt therapeutic approaches that increase performance and/ or optimize the rehabilitation process for people with changes in gait control, and patients with neurological diseases. The aim of this study is to investigate the effect of transcranial electrical stimulation (tDCS) on motor performance, autonomic control and attentional and executive functions in young individuals. A total of 20 individuals (10 women and 10 men) aged 20-30 years will participate in this study. Each participant will visit the laboratory on three occasions, interspersed for one week, one visit for the initial evaluation (approximately 1 hour) and two visits for data collection, lasting approximately 1 hour and 40 minutes each. All participants will be randomly allocated in a double-blind and counterbalanced manner in the different experimental conditions. In one of the visits will be composing the intervention group (n=10; 20 min) and in another visit the Sham group (n=10). Outcomes related to motor performance (bilateral coordination, static and dynamic balance and functional mobility), heart rate variability and attentional and executive functions will be evaluated. To this end, the gait will be analyzed through the OpenCap motion analysis system from filming and after, the phase coordination index will be calculated for analysis of bilateral coordination; the stabilometry test will be used to assess the static balance of the participants, using a force platform where the participant remains standing on the platform to measure the center of pressure; functional mobility will be investigated from the 30-second sit-up test, aiming to analyze the dynamic balance and functional strength of the lower body, and the Timed up and Go Test used for balance analysis, gait and functional capacity. Heart rate variability will be recorded from the use of the Polar Vantage heart rate monitor (Finland), with the capacity of the R-R temporal record. The attentional and executive functions will be evaluated from the Stroop Test tool. These are three tasks with 24 items each, where the participant will be evaluated according to how quickly he performs the task and the amount of errors presented. The data will be described as mean. The normality of all data will be verified by the Shapiro-Wilk test. ANOVA with repeated measures of two factors will be used, followed by the Bonferroni post hoc test to compare the variables collected between the different conditions of brain stimulation (with and without application of tDCS) and between gait conditions. One-factor ANOVA will be used for brain stimulation conditions; data will be tabulated via Excel and statistical analyses will be performed in the SPSS software package for Windows version 24.0 (IBM, Chicago, USA). A significant value of p < 0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* 20-30 years
* participant of both sex

Exclusion criteria:

* history of neurological or psychological diseases;
* use of any medications that may affect balance control, such as sedative drugs;
* presence of skeletal muscle injuries such as fracture, ligament injury, muscle tension or low back pain that restricts movement;
* presence of any sign of involvement of the spinal cord;
* visual or hearing impairment;
* musculoskeletal deformities in the lower or upper extremities that may affect the participant's standing posture;
* skin conditions (e.g., eczema and injuries) on the scalp
* presence of metal inside the head (outside the mouth) such as splinters, surgical clips or fragments of solder or metal work;
* implanted devices such as cardiac pacemaker, cochlear implant;
* score less than 24 points in the Mini Mental State Examination (MMSE)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of tDCS on motor performance | Through study completion, an average of 1 year
  * Bilateral coordination of different walking conditions will be assessed by percentage (%)
  * The static equilibrium will be evaluated by the average amplitude of displacement of the center of pressure in mean lateral and anteroposterior directions (cm)

SECONDARY OUTCOMES:
Effect of tDCS on functional mobility and dynamic balance | Through study completion, an average of 1 year
  The 30-second sit and stand test - data expressed in number of repetitions The Time Up and Go Test (TUG) - data expressed in time(s)
Effect of variability of the heart rate | Through study completion, an average of 1 year
  heart rate per min
Efect of tDCS on attentional and executive functions | Through study completion, an average of 1 year
  time (s) to realize cognitives testes (Stroob test)

CONTACTS AND LOCATIONS:
Overall Officials: Taís Malysz, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Tais Malysz, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No